CLINICAL TRIAL: NCT00439036
Title: Acceptance Therapy During Methadone Detoxification
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Angela Stotts, Associate Professor - Family Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA019436-01; R01DA019436-01 (NIH); DCNBR
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Opiate Dependence
Keywords: Opiate; Behavior Therapy; Methadone; Acceptance and Commitment Therapy (ACT)
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavior Therapy: Acceptance and Commitment Therapy (Experimental): The Act-ODT intervention consists of 24 50-minute sessions delivered weekly in the context of a methadone dose reduction program. Sessions will begin during the methadone run-up/stabilization period approximately 4 weeks prior to the onset of dose reduction and will continue through the 20 week detoxification.
  --------------------------------------------------------------------------------
  Interventions: Behavioral: Behavior Therapy
- Drug Counseling (Active Comparator): The Drug Counseling intervention consists of 24 50-minute sessions delivered weekly in the context of a methadone dose reduction program. Sessions will begin during the methadone run-up/stabilization period approximately 4 weeks prior to the onset of dose reduction and will continue through the 20 week detoxification.
  Interventions: Behavioral: Drug Counseling

INTERVENTIONS:
Behavioral: Behavior Therapy — The Act-ODT intervention will consist of 24 50-minute sessions delivered weekly in the context of a methadone dose reduction program. Sessions will begin during the methadone run-up/stabilization period approximately 4 weeks prior to the onset of dose reduction and will continue through the 20 week detoxification.
  Arms: Behavior Therapy: Acceptance and Commitment Therapy
Behavioral: Drug Counseling
  Arms: Drug Counseling

SUMMARY:
The purpose of this study is to develop an opiate detoxification behavior therapy based on current Acceptance and Commitment Therapy (ACT) theory and method, and to test its feasibility and promise in the context of voluntary methadone detoxification.

DETAILED DESCRIPTION:
This Stage I pilot study will employ a randomized, controlled, between groups design in which 70 opiate dependent patients seeking methadone detoxification will be randomized into one of two treatment conditions: ACT opiate detoxification therapy or Drug Counseling. Both therapies will be delivered in the context of a 5-month methadone dose reduction based on a linear dosing strategy. Efficacy variables will include: (1) abstinence rates during and 1-month after detoxification as assessed by regular urine screens; (2) retention of patients in treatment; and (3) patient satisfaction and treatment acceptability. Reduction in HIV/Hepatitis C risk behaviors and changes in psychosocial functioning (e.g., employment, family, legal) will also be explored, along with mediators/moderators of the therapy (i.e., experiential avoidance). Subjects will be recruited from Houston area methadone clinics and the general community via advertising and will receive methadone as part of this protocol. A 2-4 week stabilization period will precede the 5-month methadone dose reduction. During the dose reduction, participants will attend the clinic twice each week and will receive weekly therapy. Participants will be contacted for follow up assessments up to one month post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ages 25 through 60
* Dependent upon opiates (heroin/methadone) according to DSM-IV criteria
* Using heroin/methadone for at least 5 years
* Endorse 7 or higher on a 10-point motivation for opiate detoxification item
* In good physical and psychiatric health
* Able to read, speak, and understand English
* Willing and able to meet study requirements
* Willing to participate in the 1 month follow up session
* Able to provide the name of at least one person who can generally locate them
* Attending a licensed methadone clinic regularly with opiate (other than methadone) negative urine screens in the past month.
* Intake screen negative for opiates (other than methadone)
* >110 lbs & body mass index between 18 and 28 kg/m2

Exclusion Criteria:

* Younger than 25 and older than 60 years of age
* Current dependence on other substances
* Severe medical, cognitive, and/or psychiatric impairment that precludes cooperation with study protocol
* Current and severe psychiatric symptoms requiring medical attention
* Current substance withdrawal symptoms requiring medical attention
* Unable to read, speak, and understand English
* Unwillingness of women of child bearing age to use contraception
* Currently receiving other psychosocial therapy for substance abuse (12-step meetings are ok)
* Impending incarceration
* Unable or unwilling to meet study requirements, including provision of signed consent
* Less than 7 on a 10-point motivation for opiate detoxification scale
* no documentation of monitored methadone use
* non-methadone opiate positive urine screen in the past month according to self-report

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2006-07; Primary Completion 2010-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Substance use | Baseline, twice a week, end of study, one month after the study, 6 months after the study
HIV/HCV risk behaviors | Intake, week 9, week 19

SECONDARY OUTCOMES:
Retention | twice a week
Client adherence | twice a week
Psychosocial functioning | baseline and once a month
Treatment satisfaction | once a month

CONTACTS AND LOCATIONS:
Overall Officials: Angela L Stotts, Ph.D., Principal Investigator — Associate Professor- University of Texas Houston Medical School
Locations (1):
- University of Texas Medical School- Houston; Department of Psychiatry; Mental Sciences Institute, Houston, Texas, United States